CLINICAL TRIAL: NCT03355261
Title: Long-term Tracing for Axillary Lymph Nodes Dissection in the Patients With Fusion Lymph Node Before Neo-adjuvant Chemotherapy
Brief Title: Positive Node Traced Before Neoadjuvant Chemotherapy (NAC)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shengjing Hospital (Other)
Responsible Party: Principal Investigator, Jianyi Li, Principal Investigator, Shengjing Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ShengjingH01
Record Dates: First submitted 2017-11-14; First posted 2017-11-28 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Population Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- complete remission (CR) group (Experimental): According to the RECIST 1.1, 32 patients were allocated into the complete remission (CR) group based on their responses to neoadjuvant chemotherapy (NAC).
  Interventions: Procedure: complete remission (CR) group
- partial remission (PR) group (Experimental): According to the RECIST 1.1, 61 patients were allocated into the partial remission (PR) group based on their responses to neoadjuvant chemotherapy (NAC).
  Interventions: Procedure: partial remission (PR) group
- stable disease (SD) group (Experimental): According to the RECIST 1.1, 12 patients were allocated into the stable disease (SD) group based on their responses to neoadjuvant chemotherapy (NAC).
  Interventions: Procedure: stable disease (SD) group
- progressive disease (PD) group (Experimental): According to the RECIST 1.1, 5 patients were allocated into the progressive disease (PD) group based on their responses to neoadjuvant chemotherapy (NAC).
  Interventions: Procedure: progressive disease (PD) group

INTERVENTIONS:
Procedure: complete remission (CR) group — According to the RECIST 1.1, 32 patients were allocated into the complete remission (CR) group based on their responses to neoadjuvant chemotherapy (NAC).
  Arms: complete remission (CR) group
Procedure: partial remission (PR) group — According to the RECIST 1.1, 61 patients were allocated into the partial remission (PR) group based on their responses to neoadjuvant chemotherapy (NAC).
  Arms: partial remission (PR) group
Procedure: stable disease (SD) group — According to the RECIST 1.1, 12 patients were allocated into the stable disease (SD) group based on their responses to neoadjuvant chemotherapy (NAC).
  Arms: stable disease (SD) group
Procedure: progressive disease (PD) group — According to the RECIST 1.1, 5 patients were allocated into the progressive disease (PD) group based on their responses to neoadjuvant chemotherapy (NAC).
  Arms: progressive disease (PD) group

SUMMARY:
To investigate this regression model by injecting and tracing carbon nanoparticles (CNs) into the fusion node prior to NAC in patients with breast cancer.

DETAILED DESCRIPTION:
Guided by ultrasound, 0.3 mL of CNs suspension was injected in a fusion node prior to NAC in 110 patients with local advanced breast cancer. Patients underwent breast surgery and total axillary lymph node dissection following 2-6 cycles of NAC. The distribution by intercostobrachial nerves (ICBN) of positive nodes, black-stained nodes and lymphovascular invasion was investigated by response to NAC.

ELIGIBILITY:
Inclusion Criteria:

* invasive ductal carcinoma diagnosed by biopsy;
* clinically positive node diagnosed by contrast enhance computer tomography (CECT), the number of strengthened nodes at Level I ≥ 1 with the longest diameter of the strengthened node ≥ 2cm;
* NAC regimen followed the NCCN guideline;
* no prior history of breast cancer or other malignancies.

Exclusion Criteria:

* the cycle number of neo-adjuvant chemotherapy is equal to or less than 2

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2014-07-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
The spatial distribution of positive nodes in axillary after neoadjuvant chemotherapy based on pectoralis minor location | During the surgery
  After neoadjuvant chemotherapy, whether positive nodes remission (transform to negative), from Level III to Level II, and from Level II to Level I. This means that if the nodes at Level I are negative, the nodes at Level II or Level III will be negative; if the nodes at Level II are negative, the nodes at Level III will be negative; if the nodes at Level III are positive, the nodes at Level I and Level II will be positive.

SECONDARY OUTCOMES:
The spatial distribution of black-stained in axillary after neoadjuvant chemotherapy based on pectoralis minor location | During the surgery
  If the chemotherapy is sensitive, the number of black-stained nodes will increase from Level I, Level II, to Level III. If the chemotherapy is resistance, the number of black-stained nodes will remain the original number or a little increasing locally.
The spatial distribution of positive nodes in axillary after neoadjuvant chemotherapy based on intercostobrachiales nerves (ICBN) location | During the surgery
  After neoadjuvant chemotherapy, whether positive nodes remission (transform to negative), from above ICBN to below ICBN. This means that if the nodes below ICBN are negative, the nodes above ICBN will be negative; if the nodes above ICBN are positive, the nodes below ICBN will be positive.

CONTACTS AND LOCATIONS:
Overall Officials: Jianyi Li, Master, Principal Investigator — Shengjing Hospital
Locations (3):
- China (3):
  - The Second Hospital of Jilin University, Changchun, Jilin
  - the First Affiliated Hospital of China Medical University, Shenyang, Liaoning
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Li J, Jia S, Wang Y, Zhang Y, Kong L, Cao Y, Liu Y, Zhang Y, Chen B. Long-term tracing and staining of carbon nanoparticles for axillary lymph nodes in patients with locally advanced breast cancer treated with neoadjuvant chemotherapy. Asian J Surg. 2022 Jan;45(1):89-96. doi: 10.1016/j.asjsur.2021.03.020. Epub 2021 Apr 27. PMID 33926797